CLINICAL TRIAL: NCT01928095
Title: RNA Cloning and Visualization in Human Atherosclerosis
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Bradley Gelfand, PhD, Principal Investigator, University of Virginia
Other Study IDs: IRB # 13-0623-F1V
Record Dates: First submitted 2013-08-20; First posted 2013-08-23 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Atherosclerosis
Keywords: atherosclerosis; carotid endartherectomy
MeSH Terms: conditions — Atherosclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — discarded artherosclerotic tissue obtained during carotid endarterectomy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Carotid Endocardectomy Patients: Subsequent analyses will be performed on the basis of the pathological grading provided by UK Pathology (e.g do readouts of the Dicer pathway correlate with pathological plaque characteristics).

SUMMARY:
The research objectives of this project are as follows:

1. Obtain high-quality human atherosclerotic arterial samples from diseased donors.
2. Perform biochemical analysis to determine the abundance, localization and activity of Dicer and double-stranded RNAs in these diseased tissues.

DETAILED DESCRIPTION:
Participants enrolled in to this pilot study will not be randomized and will not receive any investigation medication.

In collaboration with Dr. Sibu Saha, Professor of Surgery, University of Kentucky, the investigator will obtain freshly isolated human atherosclerotic tissue from patients undergoing carotid endarterectomy. The surgical process by which the tissue is obtained is not part of this research project. These tissues are surgically removed from patients as a treatment for atherosclerosis of the carotid arteries and typically sent for pathological examination.

After the the clinical pathology has been completed, the investigator will obtain and analyze a small amount of discarded (200mg) tissue. Subsequent analyses will be performed on the basis of the pathological grading provided by UK Pathology (e.g do readouts of the Dicer pathway correlate with pathological plaque characteristics). Tissue will be anonymized, with only information with respect to drug history, age, gender and pathological grade of the tissue.

The will extract protein and RNA. Dicer abundance will be assessed by western blot, quantitative RT-PCR and northern blot. Dicer related RNAs will be measured by quantitative RT-PCR and northern blot. The invesigator will inspect the tissue for evidence of altered Dicer activity by measuring the relative levels of abundant canonical Dicer substrates/enzymatic products (i.e. the ratio of pre- to mature micro-RNA) via northern blot. The investigator predicts that Dicer levels and activity are reduced in human atherosclerotic tissue compared to healthy arteries.

Next, the investigator will assess whether downstream mediators of Dicer dysregulation are activated in these tissue samples by comparing levels and activation of the inflammasome (caspase-1, NLRP3, ASC), cytokines (IL-1β, IL-18) and signaling intermediates (MyD88, IRAK1/4) between healthy and diseased tissues. The investigator predicts that atherosclerotic plaques will exhibit evidence of Dicer dysregulation.

Next, the investigator will co-stain tissue sections with antibodies recognizing Dicer as well as cell-specific markers (CD31 for endothelium, SMA for smooth muscle, MAC-1 for macrophages) to assess whether Dicer dysregulation displays cell type-specific patterns.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 and older
* Undergoing carotid endarterectomy

Exclusion Criteria:

* Under 18 years of age
* Not undergoing carotid endarterectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and Female patients undergoing carotid endarterectomy
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2013-10; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Altered Dicer Activity | 1 year
  The investigator will measure the relative levels of abundant canonical Dicer substrates/enzymatic products (i.e. the ratio of pre- to mature micro-RNA) via northern blot

SECONDARY OUTCOMES:
Are downstream mediators of Dicer dysregulation activated | 1 Year
  Analysis will compare levels and activation of the inflammasome (caspase-1, NLRP3, ASC), cytokines (IL-1β, IL-18) and signaling intermediates (MyD88, IRAK1/4) between healthy and diseased tissues.

OTHER OUTCOMES:
Dicer dysregulation displays cell type-specific patterns. | 1 year
  The investigator will co-stain tissue sections with antibodies recognizing Dicer as well as cell-specific markers (CD31 for endothelium, SMA for smooth muscle, MAC-1 for macrophages)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Gelfand, PhD, Principal Investigator — University of Virginia, Department of Ophthalmology; Bradley Gelfand, PhD, Principal Investigator — Ophthalmology
Locations (1):
- University of Kentucky Chandler Medical Center, Lexington, Kentucky, United States